CLINICAL TRIAL: NCT04216953
Title: A Multicentre, Open-label, Phase I-II Study Evaluating the Combination of a MEK Inhibitor and a PDL1 Inhibitor in Pediatric and Adult Patients With Locally Advanced and/or Metastatic Soft Tissue Sarcoma.
Brief Title: MEK Inhibitor and a PDL1 Inhibitor Patients With Locally Advanced and/or Metastatic Soft Tissue Sarcoma
Acronym: COTESARC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET 19-036 COTESARC
Record Dates: First submitted 2019-12-18; First posted 2020-01-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Sarcoma,Soft Tissue
Keywords: MEK Inhibitor; PDL1 inhibitor
MeSH Terms: conditions — Sarcoma | interventions — cobimetinib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Cobimetinib (Experimental): Atezolimumab :
  * Adult Patient and patients ≥12 years-old with a BW ≥60kg: 840mg, Q2W
  * Pediatric Patient including patients ≥12 years-old with a BW <60kg: 15mg/kg, Q2W with a maximum of 840mg.
  Cobimetinib :
  * Pediatric patients ≥ 12 and a BW < 60kg:1mg/kg. Pediatric patients ≥ 12 and with a BW ≥ 60kg: 60mg/d.
  * Adult Patients: 60mg/d D1 to D21 over a 28-day cycle.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab

INTERVENTIONS:
Drug: Cobimetinib — Adults: 20mg film coated tablet
  Paediatrics:
  i) powder for oral suspension containing 250mg of cobimetinib
  ii) for pediatric patients ≥12 years-old and with a BW ≥60kg : 20mg film coated tablet same as adults
  Other Names: GDC-0973
Drug: Atezolizumab — 20-mL glass vial containing 1200 mg of atezolizumab.
  Other Names: RO5541267

SUMMARY:
The proposed study conducted in adult and pediatric patients aims to evaluate the safety and clinical activity of atezolizumab + cobimetinib in advanced/metastatic soft tissue sarcomas (up to 80 patients).

DETAILED DESCRIPTION:
The hypothesis of the proposed combination is as follows: cobimetinib via MEK1/2 inhibition could modify the tumor microenvironment and improve the response of T cells against tumor cells. Therefore, the addition of cobimetinib to atezolizumab may improve immune recognition and result in improved anti-tumour activity.

The combination of cobimetinib and atezolizumab showed clinical activity in a Phase I trial in patients with metastatic colorectal cancer (Atezolizumab 840 mg every 2 weeks and Cobimetinib 60 mg/d) with a disease control rate of 31%. Atezolizumab and cobimetinib are currently being tested in pediatrics in the iMatrix clinical trial with no major safety concerns to date.

A molecular screening step is mandatory for all patients enrolled in this trial in order to document MAPK pathway status and Tumor Mutational Burden (TMB) using FoundationOne test (FOne Heme).

ELIGIBILITY:
Inclusion Criteria:

I1. Male or female patients aged of at least :

- 12 years on day of signing informed consent.

I2. Histologically-confirmed diagnosis of soft tissue sarcomas, confirmed by a pathologist from RRePS Network, among the 2 cohorts:

* Rhabdomyosarcomas (RMS).
* Malign Peripheral Nerve Sheath Tumors (MPNST). I3. Availability of a representative formalin-fixed paraffin-embedded (FFPE) primary and/or metastatic tumor tissue with an associated pathology report for molecular prescreening i.e. either an archival block or a dedicated freshly collected de novo tumor biopsy.

I4. Documented MAPK pathway status and known Tumor Mutational Burden (TMB) before C1D1.

I5. Previous treatment with anthracycline-based chemotherapy (in the neoadjuvant, adjuvant or metastatic setting). Note: this criteria not mandatory for rhabdomyosarcoma.

I6. Previous treatment by at least one line of chemotherapy in the advanced/metastatic setting before C1D1.

I7. Documented radiological disease progression as per RECIST V1.1 before C1D1.

I8. At least one measurable lesion according to RECIST v1.1 before C1D1.

I9. Mandatory for adult patients only - Presence of at least one tumor lesion visible by medical imaging and accessible to repeatable percutaneous sampling that permits core needle biopsy without unacceptable risk of a significant procedural complications, and suitable for retrieval of 4 cores using a 16-gauge diameter needle or larger.

I10. Performance status:

* Karnofsky performance status for pediatric patients ≥12 years of age ≥ 70%;
* PS ECOG for adult patients: 0 or 1.

I11. Life expectancy of at least 16 weeks.

I12. Demonstrate adequate organ function based on screening laboratory tests performed within 7 days prior C1D1: Absolute neutrophil count ≥1.5 10 exp. 9/L; Platelets ≥100 10 exp. 9/L; Hemoglobin ≥9 g/dL; Serum creatinine OR Creatinine clearance according to CKD-EPI for adult and C-KID formula for pediatric patients ≤1.5 X ULN OR ≥ 30 mL/min/1.73m2 for patient with creatinine levels > 1.5 ULN; Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN; ASAT and ALAT and ALP ≤ 3 X ULN; INR and Activated Partial Thromboplastin Time (aPTT)≤1.5 X ULN; Troponin T or I negative (< ULN).

I13. Resolution (i.e. ≤ Grade 1 with the exception of alopecia all grades and Grade 2 for neuropathy, lab values presented in criteria I12.) of any toxicities related to previous anti-cancer treatment.

I14. Women patient of child-bearing potential must have a negative serum pregnancy test before C1D1 and must agree to use effective forms of contraception from the time of the negative pregnancy test up to 6 months after the last dose of study drugs.

I15. Sexually active and fertile men must agree to use contraceptive measures up to 5 months after the last study drugs.

I16. Written informed consent from patient, parents if applicable/legal representative, before any study-specific screening procedures, and willingness to comply to study visits and procedures.

I17. Patients must be covered by a medical insurance.

Exclusion Criteria:

NI1. Soft tissue sarcoma disease considered curable with surgery or radiotherapy.

NI2. Prior treatment with cobimetinib or other MEK inhibitors. NI3. Prior treatment with immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, or anti-PD-L1 therapeutic antibodies.

NI4. Patients with history of severe allergic or other hypersensitivity reactions to:

* Chimeric or humanized antibodies or fusion proteins,
* Biopharmaceuticals produced in Chinese hamster ovary cells, or
* Any component of the atezolizumab formulation.
* Any component of Cobimetinib formulation.

NI5. History of malabsorption syndrome or other condition that would interfere with the absorption of oral medications.

NI6. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

Note: Asymptomatic patients with treated CNS lesions are eligible, provided that all of the following criteria are met:

* Measurable disease, per RECIST v1.1, must be present outside the CNS.
* No history of intracranial hemorrhage or spinal cord hemorrhage.
* Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
* No stereotactic radiotherapy within 7 days prior to initiation of study treatments, whole-brain radiotherapy within 14 days prior to initiation of study treatment, neurosurgical resection within 28 days prior to initiation of study treatments.
* No evidence of interim progression between completion of CNS-directed therapy and initiation of study treatments.
* No ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted.

NI7. History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, central serous chorioretinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration.

NI8. Left ventricular ejection fraction (LVEF) < institutional lower limit of normal (according to age) or < 50%.

NI9. History of congenital long QT syndrome or corrected QT interval (QTc) > 450 ms.

NI10. Patients using, or requirement to use while on the study, or not respecting the minimal wash-out period of medications listed below:

Any approved anti-cancer systemic treatment including chemotherapy, hormonotherapy, biological therapy, or immunotherapy: 2 weeks; any investigational agents: 4 weeks; Radiotherapy: 3 weeks; major surgical procedure, open biopsy, or significant traumatic injury: 4 weeks; abdominal surgery, abdominal interventions or significant abdominal traumatic injury : 60 days; live vaccines : 4 weeks; systemic immunostimulatory agents, including but not limited to IFN-α, IFN-γ, or IL-2 : 4 weeks; immunosuppressive medications with the exceptions of intranasal, inhaled, or topical corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid: 2 weeks; P-gp inhibitors : None; Strong or moderate inhibitors of CYP3A4 : None; Strong CYP3A4 inducers: None; oral or IV antibiotics : 2 weeks.

NI11. Patients with a malignancy other than STS within 5 years prior to C1D1 with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome

NI12. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis with the following exceptions:

* patients with a history of autoimmune-related hypothyroidism who are on stable thyroid replacement hormone therapy,
* patients with controlled Type 1 diabetes mellitus,
* patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are eligible provided that they meet the following conditions:
* rash must cover less than 10% of body surface area (BSA).
* disease is well controlled at baseline and only requiring low potency topical steroids.
* no acute exacerbations of underlying condition within the previous 12 months requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids.

NI13. Patients with HIV, active B or C hepatitis infection, or any other active infection.

Active hepatitis C i.e. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA at screening.

NI14. Patients with active tuberculosis. NI15. Prior allogeneic bone marrow transplantation or solid organ transplant for another malignancy in the past.

NI16. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan.

NI17. Patients with a high-risk of hemorrhage or history of coagulopathy. NI18. Pregnant or breastfeeding women. N19. Patients with a history of immune-mediated pericardial disorder (including pericarditis) related to immune-stimulatory anticancer agents

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Phase II part | 16 weeks
  The Progression Free rate after 16 weeks of treatment is defined as the rate of patients with a complete response or a partial response or a stable disease as per RECIST V1.1.

SECONDARY OUTCOMES:
Objective response rate | at 8 weeks and 16 weeks
  The objective response rate at 8 (16) weeks is defined as the proportion of patients with a complete response or a partial response after 8 (16) weeks of treatment.
Duration of response | Time interval from the date of first occurrence of a documented objective response until the date of documented progression or death in the absence of disease progression up to 3 month.
  Duration of response is defined as the time interval from the date of first occurrence of a documented objective response (CR or PR, whichever status is recorded first) until the date of documented progression or death in the absence of disease progression.
Progression-free survival | Time from the first day of study treatment to the date of the first documented tumor progression or death up to 3 month.
  Progression-free survival (PFS) is defined as the time from the first day of study treatment to the date of the first documented tumor progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Nadège Corradini, MD, Principal Investigator — Centre Leon Berard
Locations (6):
- France (6):
  - Institut de Cancérologie de l'Ouest, Angers
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif